CLINICAL TRIAL: NCT01427387
Title: Phase I Study of ASP0456 - A Double-blind, Placebo-controlled, Multiple Ascending Dose Study / Investigational Study for Dose Timing Selection in Non Elderly Healthy Subjects-
Brief Title: A Study to Evaluate Safety of Multiple Dose of ASP0456 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 0456-CL-0012
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Healthy; Pharmacokinetics of ASP0456
Keywords: ASP0456; Pharmacokinetics; safety; tolerability; food effect
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part-1 ASP group (Experimental): ASP0456 receiving group
  Interventions: Drug: ASP0456
- Part-1 Placebo group (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo
- Part-2 group (Experimental): cross-over study group to evaluate food effect on ASP0456 plasma concentration
  Interventions: Drug: ASP0456

INTERVENTIONS:
Drug: ASP0456 — oral
  Other Names: linaclotide
  Arms: Part-1 ASP group; Part-2 group
Drug: Placebo — oral
  Arms: Part-1 Placebo group

SUMMARY:
A study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending dose of ASP0456 in non-elderly healthy subjects. Two dosing condition, pre-prandial and postprandial administrations, is compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as judged by the investigator/subinvestigator based on the results of physical examination and all tests obtained
* Body weight (at screening);

  * female ≥40.0 kg,<70.0 kg
  * male ≥50.0 kg,<80.0 kg
* BMI(at screening): ≥17.6,<26.4

Exclusion Criteria:

* Received any investigational drugs in other clinical or post-marketing studies within 120 days before the study
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before the study
* Received medication within 10 days before dose is administered or is scheduled to receive medication
* History of drug allergies
* Upper (e.g. nausea, vomiting, stomachache) and lower (e.g. abdominal pain) gastrointestinal disease within 7 days before the study
* Concurrent or previous hepatic disease
* Concurrent or previous heart disease
* Concurrent or previous renal disease

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (such as Cmax, AUC and t1/2 etc.) of ASP0456 assessed by its plasma concentration change | For 48 hours after dosing

SECONDARY OUTCOMES:
Safety assessed by the incidence of adverse events, vital signs, 12-lead ECGs and labo tests | For 48 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Use Cental Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan